CLINICAL TRIAL: NCT04375332
Title: A Prospective, Multi-center Trial to Evaluate the Safety and Effectiveness of Beating Heart Mitral Valve Repair With the HARPOON™ System (RESTORE)
Brief Title: Beating Heart Mitral Valve Repair With the HARPOON™ System
Acronym: RESTORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HARPOON™ Beating Heart Mitral Valve Repair System (Experimental): Subjects who were treated with the HARPOON™ Beating Heart Mitral Valve Repair System
  Interventions: Device: HARPOON™ Beating Heart Mitral Valve Repair System

INTERVENTIONS:
Device: HARPOON™ Beating Heart Mitral Valve Repair System — Repair of the chordae tendinae in the mitral valve.

SUMMARY:
The objective of the study is to evaluate the safety and effectiveness of the HARPOON™ System in the treatment of patients with severe degenerative mitral regurgitation (DMR).

DETAILED DESCRIPTION:
RESTORE is a prospective, multicenter, non-randomized trial designed to evaluate the safety and effectiveness of the HARPOON™ Beating Heart Mitral Valve Repair System in patients with severe degenerative mitral regurgitation (DMR).

ELIGIBILITY:
Inclusion Criteria:

Each subject is required to meet all of the following inclusion criteria:

1. Patient is >/= 21 years old.
2. Presence of severe degenerative mitral regurgitation with mid-segment posterior leaflet prolapse (without commissural involvement) by echocardiographic study.
3. Mitral leaflet coaptation surface sufficient to reduce mitral regurgitation without undue leaflet tension, based on the judgment of the Echocardiographic Core Lab.
4. Patient competent to sign informed consent and able to return for follow-up and is capable of participating in all testing associated with this clinical investigation.

Exclusion Criteria:

Patients will be excluded if ANY of the following criteria apply:

1. Functional mitral regurgitation (FMR).
2. Evidence of anterior or bileaflet prolapse.
3. Severe mitral annular calcification (MAC).
4. Moderate or greater leaflet calcification.
5. Fragile or thinning apex (e.g. LV aneurysm).
6. Have undergone cardiac or peripheral vascular procedures within 30 days prior to the trial procedure.
7. Planned cardiac or peripheral vascular procedures within 30 days after the trial procedure.
8. Requirement for concomitant cardiac surgery.
9. Severe pulmonary hypertension (pulmonary artery systolic pressure > 60mmHg).
10. Severe aortic stenosis or insufficiency.
11. Severe tricuspid regurgitation. (Patients with mild or moderate tricuspid regurgitation are not excluded.)
12. Left ventricular ejection fraction (LVEF) <30%, or severely impaired right ventricular dysfunction as measured by the core lab.
13. Any history of endocarditis.
14. Contraindication to cardiac surgery, including hostile chest or history of mediastinal radiation.
15. Previous structural heart intervention (e.g. any heart valve replacement or repair procedures). Previous percutaneous coronary intervention (PCI) is allowed.
16. Previous coronary artery bypass grafting (CABG).
17. Stroke within 30 days prior to index procedure.
18. ST segment elevation myocardial infarction (STEMI) requiring intervention within 30 days prior to index procedure.
19. Evidence of cirrhosis or hepatic synthetic failure (Child-Pugh Class B or higher, [or MELD score of ≥ 13]).
20. Renal insufficiency CKD Stage 3b or worse (GFR < 45 ml/min/1.73 m2).
21. Hemodynamic instability or cardiogenic shock at the time of enrollment (e.g. requiring inotropic support or mechanical support devices).
22. History of bleeding diathesis or coagulopathy or leukopenia (WBC < 3000 mcL) or acute anemia (Hb < 9 g/dL) or thrombocytopenia (platelets < 50,000 cells mcL).
23. Active SARS-CoV-2 infection (Coronavirus-19 [COVID-19]) or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments (as assessed by Case Review Committee).
24. Refuse blood products.
25. Planned treatment with any other investigational device or procedure through 1-year follow-up, or who are currently participating in an investigational drug or device trial.
26. Carotid stenosis ≥ to 80% at time of enrollment.
27. Rheumatic heart disease including rheumatic mitral stenosis.
28. Pregnant or lactating at the time of enrollment (women of childbearing age should have negative pregnancy test within 72 hours of surgery) or planning pregnancy within the next 12 months.
29. Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator.
30. Condition or conditions that, in the opinion of the Investigator, precludes participation, including willingness to comply with all follow-up procedures.
31. Contraindication for transesophageal echocardiography (TEE), including esophageal spasm, esophageal stricture, esophageal laceration, esophageal perforation, esophageal diverticula (e.g. Zenker's diverticulum).
32. Echocardiographic evidence of intracardiac mass (e.g. left ventricular, atrial, or appendage thrombus, myxoma, or vegetation).
33. Cannot tolerate procedural anticoagulation or post-procedure antiplatelet regimen.

    Intra-operative exclusion criteria
34. No longer meets eligibility criteria based on intra-operative assessment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in NYHA classification from Baseline to 5 years | Baseline compared to 1 and 5 years
  The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life. Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Symptoms of heart failure or the anginal syndrome may be present even at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod H. Thourani, MD, Principal Investigator — Dept of Cardiovascular Surgery, Piedmont Heart Institute; Konstantinos Koulogiannis, MD, Principal Investigator — Department of Cardiovascular Medicine Gagnon Cardiovascular Institute
Locations (9):
- United States (9):
  - UCSF, San Francisco, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - OHSU Knight Cardiovascular Institute, Portland, Oregon
  - Centennial Medical Center, Nashville, Tennessee
  - Intermountain Heart Institute, Murray, Utah

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.